CLINICAL TRIAL: NCT02260596
Title: A Multicenter Consortium to Define the Epidemiology and Outcomes of Respiratory Viral Infections in Pediatric Transplant Recipients
Brief Title: Respiratory Viral Infections in Pediatric Transplantation
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Washington (Other); Children's Hospital of Philadelphia (Other); Albert Einstein College of Medicine (Other); Baylor College of Medicine (Other); St. Jude Children's Research Hospital (Other); University of Cincinnati (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00056727
Record Dates: First submitted 2014-09-29; First posted 2014-10-09 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-07

CONDITIONS: Infection in Solid Organ Transplant Recipients; Complications of Organ Transplant; Respiratory Viral Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort Population: Pediatric SOT/HSCT recipients

SUMMARY:
A retrospective cohort of solid organ transplant (SOT) and hematopoietic stem cell transplant (HSCT) recipients will be assembled to determine the incidence of respiratory viral infections diagnosed during an inpatient admission in the first year post-transplant. A sub-cohort of patients that develop a respiratory viral infection within one year of transplantation will be leveraged to investigate factors associated with mortality in the three months after respiratory viral infection.

DETAILED DESCRIPTION:
The purpose of the study is to 1) Determine the incidence of respiratory viral infections diagnosed during the first year post SOT and HSCT; 2a) Determine the all-cause mortality within 3 months of a respiratory viral infection diagnosed during an inpatient admission in the first year post SOT and HSCT; 2b) Determine the proportion of deaths within 3 months of a respiratory viral infection diagnosed during an inpatient admission deemed to be directly attributable to that infection; and 3) To identify factors known at time of onset of the inpatient respiratory viral infection that are associated with all-cause mortality. The study cohort will consist of any SOT or HSCT recipient ≤18 years of age that received their transplant between January 1st, 2010 and June 30th, 2013. Th cohort will determine the incidence of respiratory viral infections diagnosed during an inpatient admission in the first year post-transplant. A sub-cohort of patients that develop a respiratory viral infection within one year of transplantation will be leveraged to investigate factors associated with mortality in the 3 months after respiratory viral infection. Baseline and demographic characteristics will be summarized by standard descriptive summaries. Categorical variables will be summarized by frequencies while continuous variables will be summarized using mean, standard deviation and/or median, twenty-fifth and seventy-fifth percentiles, minimum, and maximum. This is a minimal risk study using data that will be collected retrospectively from medical charts. The only potential risk would be loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 0 to <18 years at the time of HSCT or SOT
* Transplantation occurred between January 1st, 2010 and June 30th, 2013.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study cohort will consist of any SOT or HSCT recipient ≤18 years of age that received their transplant between January 1st, 2010 and June 30th, 2013. Participants will have information collected from 30 days prior to transplant until the first of the following: 365 days post receipt of transplant, death, or loss to follow-up. If a patient has more than one viral respiratory infection of the same pathogen during the study period, then only the first infection will be considered unless isolated at least one month after the first positive test and only if after at least two negative tests for that same virus. A patient can contribute more than one viral respiratory infection if they are caused by different viral pathogens.
Sampling Method: Non-Probability Sample
Enrollment: 2669 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory viral infection | 1 year post transplant
  Pediatric SOT/HSCT recipients who do not develop respiratory viral infection within 1 year following transplant

SECONDARY OUTCOMES:
All-cause mortality of respiratory viral infection | 3 months after respiratory viral infection
  Determine the all-cause mortality within 3 months of a respiratory viral infection diagnosed during an inpatient admission in the first year post SOT and HSCT.

OTHER OUTCOMES:
Factors associated with all-cause mortality of respiratory viral infection | 3 months after respiratory viral infection
  This tertiary aim will include just those patients that had an inpatient respiratory viral infection. The analysis will explore the association of factors known at time of onset of the respiratory viral infection with 3 month all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: William J Steinbach, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States